CLINICAL TRIAL: NCT00751595
Title: A Phase II Randomized, Open Label, Immunogenicity and Safety Trial of the Vaccine Based on the Recombinant Biologically Active HIV-1 Tat Protein in Anti-Tat Negative HIV-1 Infected HAART-treated Adult Subjects.
Brief Title: Immunogenicity and Safety Trial of the HIV-1 Tat Vaccine
Acronym: ISS T-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ensoli, MD (Other)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PHD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISS T-002
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: HIV; Tat protein; Therapeutic vaccine; HAART; HIV Therapeutic Vaccine; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Gene Products, tat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Tat Protein 7.5 or 30 microg 5X) (Experimental): Group I: Subjects receiving 5 intradermal immunization with Tat (7.5 microg); Group II: Subjects receiving 5 intradermal immunization with Tat (30 microg).
  Interventions: Biological: Tat protein
- ARM B (Tat Protein 7.5 or 30 microg, 3X) (Experimental): Group I: Subjects receiving 3 intradermal immunization with Tat (7.5 microg); Group II: Subjects receiving 3 intradermal immunization with Tat (30 microg)
  Interventions: Biological: Tat protein

INTERVENTIONS:
Biological: Tat protein — Biologically active recombinant Tat protein

SUMMARY:
The study is a randomized, open label, phase II clinical trial directed at evaluating the immunogenicity (as a primary end-point) and the safety (as a secondary end-point), of the recombinant HIV-1 Tat vaccine in HIV-1 infected adult subjects, anti-Tat antibody negative, HAART-treated with chronic suppressed HIV-1 infection, CD4+ T cell counts >= 200 cells/microliter, levels of plasma viremia < 50 copies/ml in the last 6 months prior to the screening and without a history of virologic rebound. The immunogenicity of 3 or 5 immunizations of the two different vaccine doses (7.5 and 30 micrograms) of the Tat vaccine has been evaluated.

DETAILED DESCRIPTION:
This phase II clinical trial was directed at evaluating the immunogenicity and the safety of the HIV-1 Tat protein-based vaccine. Anti-Tat antibody negative, HIV-1 positive subjects treated successfully with HAART have been screened and recruited for a 48-weeks study, including a period of 16 or 8 weeks treatment phase and a period of 32 or 40 weeks follow-up phase, in arm A or Arm B, respectively. One hundred sixty-eight subjects have been randomized 1:1:1:1 to one of the 2 arms (Arm A and Arm B) and each arm has been divided in the following groups:

Arm A - Group I: 5 immunizations with Tat (7.5 microg) at weeks 0, 4, 8, 12, 16; Arm A - Group II: 5 immunizations with Tat (30 microg) at weeks 0, 4, 8, 12, 16; Arm B - Group I: 3 immunizations with Tat (7.5 microg) at weeks 0, 4, 8; Arm B - Group II: 3 immunizations with Tat (30 microg) at weeks 0, 4, 8.

Four vaccination regimens have been tested by intradermal administration of the Tat vaccine at two different doses (7.5 microg or 30 microg) in 5 or 3 immunizations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Anti-Tat antibody negative subjects
* HIV-1 infected subjects under successful HAART treatment with HIV plasma viremia < 50 copies/ml in the last 6 months prior to the screening
* Subjects with any pre-HAART CD4 nadir;
* CD4+ T cell counts ≥ 200 cells/μl at enrolment;
* Availability for the planned study duration
* Negative pregnancy test for women of childbearing potential (to be performed during the screening phase and just before the immunizations) and use of an acceptable mean of contraception (condom, hormonal or mechanical methods) for one month prior to immunization and for the all duration of the study
* Signed informed consent

Exclusion Criteria:

* Concomitant AIDS-related opportunistic disease;
* Concomitant neoplastic diseases;
* History of malignant neoplastic diseases [NOTE: Subjects with history of non malignant neoplastic diseases completely resolved according to the fulfillment of all the specific recovery criteria, in agreement with the current guidelines in medical oncology are eligible];
* History of encephalopathy, neuropathy or unstable CNS pathology, immunodeficiency, autoimmune disease, angina or cardiac arrhythmias, or any other clinically significant medical problems;
* Any evidence, as judged by the investigator, of unstable cardio-vascular disease (e.g. unstable hypertensive disease needing modification or introduction of an anti-hypertensive treatment);
* Chest radiography showing evidence of active or acute cardiac or pulmonary disease within 6 months prior to study screening visit;
* History of anaphylaxis or serious adverse reactions to vaccines as well as serum IgE levels exceeding 1000 U.I./ml;
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g. Steven-Johnson syndrome, bronchospasm, or hypotension);
* Active tuberculosis documented PPD skin test within one year [NOTE: if the PPD skin test is positive, then a chest x-ray will be done and if no findings consistent with active pulmonary tuberculosis and no indications exist for prophylaxis or treatment, the subject is eligible for participation in this trial];
* Medical or psychiatric condition which preclude subject compliance with the protocol. Specifically, persons with psychotic disorders, major affective disorders, suicidal ideation are to be excluded;
* Current use of psychotropic drugs prescribed for major psychotic disorders;
* Concomitant participation in any experimental study;
* Current or prior therapy with immunomodulators or immunosuppressive drugs and anticoagulant drugs within 30 days prior to study medication administration;
* Live attenuated vaccines within 60 days of study inclusion [NOTE: Medically indicated sub-unit or killed vaccines (e.g., influenza, pneumococcal, hepatitis A and B) are not exclusionary, but should be given at least 4 weeks away from HIV immunizations];
* Receipt of blood products or immunoglobulin in the past year;
* Previous participation in an HIV-1 vaccine trial (subjects who despite their participation as placebo in a HIV-1 vaccine trial have never been effectively administered with a HIV-1 vaccine are eligible);
* Drug and/or alcohol abuse;
* Use in the last 6 months or concomitant use of anti CCR5 inhibitors and/or integrase inhibitors and/or fusion inhibitors;
* Pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Humoral and cellular immune responses to Tat | up to 144 weeks
  It has been measured by the induction, magnitude and persistence of the humoral and cellular immune responses to Tat and by comparing the immunogenicity of a 3 or 5 immunizations of the 7.5 microg and 30 microg vaccine doses.

SECONDARY OUTCOMES:
The Secondary Endpoint has been focused on adverse events, including any significant change in hematological/biochemical and coagulation laboratory parameters. | up to 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ensoli, MD, PhD, Study Director — National AIDS Center (CNAIDS), Istituto Superiore di Sanita', Rome, Italy
Locations (11):
- Italy (11):
  - San Gerardo Hospital, Monza, Milan
  - General Hospital of Bari, Bari
  - Spedali Civili di Brescia, Brescia
  - General Hospital-University of Ferrara, Ferrara
  - A.M. Annunziata Hospital, Florence
  - S.M. Goretti Hospital, Latina
  - San Raffaele Hospital, Milan
  - L. Sacco Hospital, Milan
  - General Hospital-University of Modena, Modena
  - San Gallicano Hospital, Rome
  - Amedeo di Savoia Hospital, Torino

REFERENCES:
- [Background] Butto S, Fiorelli V, Tripiciano A, Ruiz-Alvarez MJ, Scoglio A, Ensoli F, Ciccozzi M, Collacchi B, Sabbatucci M, Cafaro A, Guzman CA, Borsetti A, Caputo A, Vardas E, Colvin M, Lukwiya M, Rezza G, Ensoli B; Tat Multicentric Study Group. Sequence conservation and antibody cross-recognition of clade B human immunodeficiency virus (HIV) type 1 Tat protein in HIV-1-infected Italians, Ugandans, and South Africans. J Infect Dis. 2003 Oct 15;188(8):1171-80. doi: 10.1086/378412. Epub 2003 Sep 30. PMID 14551888
- [Background] Cafaro A, Caputo A, Maggiorella MT, Baroncelli S, Fracasso C, Pace M, Borsetti A, Sernicola L, Negri DR, Ten Haaft P, Betti M, Michelini Z, Macchia I, Fanales-Belasio E, Belli R, Corrias F, Butto S, Verani P, Titti F, Ensoli B. SHIV89.6P pathogenicity in cynomolgus monkeys and control of viral replication and disease onset by human immunodeficiency virus type 1 Tat vaccine. J Med Primatol. 2000 Aug;29(3-4):193-208. doi: 10.1034/j.1600-0684.2000.290313.x. PMID 11085582
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Monini P, Magnani M, Garaci E. The therapeutic phase I trial of the recombinant native HIV-1 Tat protein. AIDS. 2008 Oct 18;22(16):2207-9. doi: 10.1097/QAD.0b013e32831392d4. PMID 18832884
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- [Background] Bellino S, Francavilla V, Longo O, Tripiciano A, Paniccia G, Arancio A, Fiorelli V, Scoglio A, Collacchi B, Campagna M, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Parallel conduction of the phase I preventive and therapeutic trials based on the Tat vaccine candidate. Rev Recent Clin Trials. 2009 Sep;4(3):195-204. doi: 10.2174/157488709789957529. PMID 20028332
- [Background] Longo O, Tripiciano A, Fiorelli V, Bellino S, Scoglio A, Collacchi B, Alvarez MJ, Francavilla V, Arancio A, Paniccia G, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Phase I therapeutic trial of the HIV-1 Tat protein and long term follow-up. Vaccine. 2009 May 26;27(25-26):3306-12. doi: 10.1016/j.vaccine.2009.01.090. Epub 2009 Feb 7. PMID 19208456
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Result] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Result] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Result] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Result] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- See also: Related Info — http://www.hiv1tat-vaccines.info